CLINICAL TRIAL: NCT01444599
Title: Virtual Histology (VH)-Intravascular Ultrasound (IVUS) Tissue Characteristics Analysis of the Intermediate Coronary Artery Stenosis Lesion Predicting Physiologic Myocardial Ischemia by Myocardial Fraction Flow Reserve (FFR)
Brief Title: VH-IVUS Plaque Composition Analysis By Fractional Flow Reserve
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Joon Hyung Doh, Associate Professor of Medicine, Inje University
Other Study IDs: IB-1110-048
Record Dates: First submitted 2011-09-26; First posted 2011-10-03 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Disease
Keywords: coronary atherosclerosis; virtual histology intravascular ultrasound; fractional flow reserve
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- low FFR group (<0.8): the patient with FFR values less than 0.8
- high FFR group (>0.8): the patient with FFR values greater than 0.8

SUMMARY:
Recent clinical trials demonstrated that virtual histology-intravascular ultrasound (VH-IVUS) is a useful test predicting clinical outcomes of the coronary artery disease (CAD). Thin cap fibroatheroma (VH-TCFA) was proposed a predictor of cardiovascular event by VH-IVUS combined with more than 70% plaque burden and less than 4mm² minimal lumen area (MLA) by IVUS. Fractional flow reserve (FFR) is an established index of the physiological significance of a coronary stenosis. Recent large scale trials demonstrated FFR guided PCI showed favorable clinical outcomes. VH-IVUS represents anatomical severity, but FFR represents functional severity of CAD. Few studies reported relevance between two tests. Aim of this study was to investigate whether the geometry and composition of lesions were different under FFR criteria.

ELIGIBILITY:
Inclusion Criteria:

* clinical angina pectoris who underwent VH-IVUS and FFR during coronary angiography.
* agree with informed consent

Exclusion Criteria:

* unable to get informed consent
* low left ventricular ejection fraction less than 35%
* chronic renal failure (Cr>2.0mg/dl)
* acute myocardial infarction related coronary artery
* allergy to adenosine injection

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent coronary angiography for the diagnostic purposes because of clinical angina pectoris. Patient who underwent simultaneous virtual histology-intravascular ultrasound (VH-IVUS)and fractional flow reserve (FFR) measurement at the time of coronary angiography would be enrolled consecutively.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-03; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Differences VH-IVUS plaque composition between different FFR groups | baseline
  VH-IVUS tissue composition (necrotic core, dense calicium, fibrotic, fibrofatty %) and atheroma type will be compared according to different FFR groups at the time of measurement procedure.

SECONDARY OUTCOMES:
Serial physiologic and plaque composition changes of deferred lesions at 1 year FFR and VH-IVUS follow-up. | one year
  Approximately 60-70 of 100 enrolled patients would be deferred according to FFR values. Patient who provide consent for clinical and angiographic follow-up at one year would be assessed by physiologic FFR and VH-IVUS derived plaque composition. Relationship of serial physiologic and plaque composition changes will be evaluated. Anatomic and physiologic parameters associated with plaque progression and/or regression will be determined.
Serial physiologic and plaque composition changes of stented lesions at 1 year FFR and VH-IVUS follow-up. | one year
  Approximately 30-40 of 100 enrolled patients would be stented according to FFR values. Patient who provide consent for clinical and angiographic follow-up at one year would be assessed by physiologic FFR and VH-IVUS derived plaque composition including stented segment. Relationship of serial physiologic and plaque composition changes will be evaluated. Anatomic and physiologic parameters associated with stent failure will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Joon Hyung Doh, MDPhD, Principal Investigator — Inje University Ilsan Paik Hospital
Locations (4):
- South Korea (4):
  - Inje University Ilsan Paik Hospital, Goyang, Gyeonggido
  - Seoul National University Hospital, Seoul, Seoul
  - Keimyung University Dongsan Medical Center, Daegu
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Background] Brugaletta S, Garcia-Garcia HM, Shen ZJ, Gomez-Lara J, Diletti R, Sarno G, Gonzalo N, Wijns W, de Bruyne B, Alfonso F, Serruys PW. Morphology of coronary artery lesions assessed by virtual histology intravascular ultrasound tissue characterization and fractional flow reserve. Int J Cardiovasc Imaging. 2012 Feb;28(2):221-8. doi: 10.1007/s10554-011-9816-3. Epub 2011 Feb 19. PMID 21336551
- [Background] Kubo T, Maehara A, Mintz GS, Doi H, Tsujita K, Choi SY, Katoh O, Nasu K, Koenig A, Pieper M, Rogers JH, Wijns W, Bose D, Margolis MP, Moses JW, Stone GW, Leon MB. The dynamic nature of coronary artery lesion morphology assessed by serial virtual histology intravascular ultrasound tissue characterization. J Am Coll Cardiol. 2010 Apr 13;55(15):1590-7. doi: 10.1016/j.jacc.2009.07.078. PMID 20378076
- [Background] Stone GW, Maehara A, Lansky AJ, de Bruyne B, Cristea E, Mintz GS, Mehran R, McPherson J, Farhat N, Marso SP, Parise H, Templin B, White R, Zhang Z, Serruys PW; PROSPECT Investigators. A prospective natural-history study of coronary atherosclerosis. N Engl J Med. 2011 Jan 20;364(3):226-35. doi: 10.1056/NEJMoa1002358. PMID 21247313